CLINICAL TRIAL: NCT03419390
Title: A Prospective,Open Label,Non-randomized,Single-centre,Exploratory,Stratified Pilot Study for the Evaluation of the Safety and Performance of a Combined Coaxial Optical Coherence Tomography (OCT) System,to Image Diseases of the Posterior and Anterior Segment of the Eye
Brief Title: A Pilot Study for the Evaluation of the Safety and Performance of a Combined OCT System
Acronym: Hydra01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 085-HAP-2017-001
Record Dates: First submitted 2017-11-17; First posted 2018-02-05 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Healthy
Keywords: Hydra01
MeSH Terms: interventions — Tomography, Optical Coherence; Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Proof of concept study, medical device investigation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy subjects (Other): One eye of each participant will be scanned with the investigational device (= combined Coaxial Optical Coherence Tomography (OCT) System)
  Interventions: Device: combined Coaxial Optical Coherence Tomography (OCT) System
- Diseased groups (Other): lf one eye is affected, this will be chosen. lf both eyes are be affected, the eye with the severest symptoms will be chosen. Scanning with the investigational device (= combined Coaxial Optical Coherence Tomography (OCT) System)
  Interventions: Device: combined Coaxial Optical Coherence Tomography (OCT) System
- Diseased subgroups (Other): Every second subject will be allocated to the subgroup.
  1. Scanning with the investigational device (= combined Coaxial Optical Coherence Tomography (OCT) System)
  2. Thickness measurement with reference medical device.
  Interventions: Device: combined Coaxial Optical Coherence Tomography (OCT) System

INTERVENTIONS:
Device: combined Coaxial Optical Coherence Tomography (OCT) System — The investigational device is an OCT scanner prototype with two different wavelengths developed based on a CE marked OCT device (Spectralis® Heidelberg) at the Berner Fachhochschule, Biel

SUMMARY:
The novel Coaxial Optical Coherence Tomography (OCT) System is designed to visualize both structures of the retina and choroid.

The purpose of this research is the safety and evaluation of a combined coaxial optical coherence tomography (OCT) system, to image diseases of the posterior and anterior segment of the eye.

DETAILED DESCRIPTION:
Background and Rationale:

Many posterior segment ocular diseases involve the retinal and choroidal vasculature. A new technology to noninvasively and simultaneously visualize vascular pathology is of utmost importance to reduce patient exposure to different diagnosis methods like e.g. fluorescence angiography. The novel Coaxial Optical Coherence Tomography (OCT) System is designed to visualize both structures of the retina and choroid.

Furthermore, it may be used to image other structures of the eye.

Objective(s):

The purpose of this research is the safety and evaluation of a combined coaxial optical coherence tomography (OCT) system, to image diseases of the posterior and anterior segment of the eye. This device may be useful for the early diagnosis and monitoring of a variety of diseases involving the eye, such as Glaucoma, Diabetic Retinopathy or Age-Related Macular Degeneration. Measurements are compared to normal controls.

Measurements and procedures:

After screening, all participants will undergo a scanning procedure on the same day.

Only one eye of each participant will be scanned with the investigational device. For patients, the eye showing the disease will be chosen, for healthy volunteers, the left or right eye will be scanned according to a randomisation list.

The image quality is rated by the investigator and an independent assessor on a VAS (visual analogue scale). A subgroup of each stratum will have a comparative measurement of the choroid thickness against a SS-OCT (swept-source-OCT) device (Topcon) and a retina thickness against the Spectralis data. The subgroup will consist of half planned sample size. The measurement is taken from one eye, ie. every second participant per stratum will be attributed to the thickness measurement subgroup. The endpoint is a true/false criterion on whether the measurement of the retina and choroid thickness was successful. The thickness is measured in μm. The measurement is considered a "success" if the value is no more than +/- 10% off the reference measurement.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with healthy eye, or has been diagnosed already with eye disease
* Patients > 18 years of age
* Informed Consent as documented by date and signature

Exclusion Criteria:

* Clinically significant concomitant disease that impair measurement
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, late stage Alzheimer disease, etc. of the participant,
* Subjects using implanted electronic medical devices (e.g. cochlear implant, pacemaker, defibrillator, infusion pump).
* Participation in another study with investigational drug within the 30 days preceding and during the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Visual acuity (VA) after investigation | Within 1 hour after investigation
  Safety of the imaging investigation expressed as visual acuity before (baseline) and after imaging, and tolerability assessment questionnaire.

SECONDARY OUTCOMES:
Scan quality | After completion of all measurement, an average of 2 years.
  Comparing scan quality of investigational device to scan quality of a reference device, expressed as thickness of the retina and the thickness of the choroid
Procedural success | After completion of all measurement, an average of 2 years.
  Procedural success that is defined as: Image Quality of anterior and posterior eye structures
Procedural safety and comfort assessed by questionnaire | Within 1 hour after investigation
  Procedural comfort in the opinion of the patients assessed with a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik PN Scholl, MD, Study Director — University Hospital Basel, Dept. of Ophthalmology; Pascal Hasler, MD, Principal Investigator — University Hospital Basel, Dept. of Ophthalmology